CLINICAL TRIAL: NCT00903630
Title: Phase I/II Trial of Lenalidomide in Combination With Liposomal Doxorubicin for the Treatment of Recurrent Epithelial Ovarian, Fallopian Tube and Primary Peritoneal Cancer
Brief Title: Lenalidomide and Doxorubicin Hydrochloride Liposome in Recurrent Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008LS047; 0805M32463 (Other: IRB, University of Minnesota); WCC #50 (Other: Women's Cancer Center, University of Minnesota); RV-OVAR-PI-0447 (Other: Celgene Corporation)
Record Dates: First submitted 2009-05-15; First posted 2009-05-18 (Estimated); Results first posted 2017-01-18 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; fallopian tube cancer; peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Lenalidomide; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase 1 - Dose Level 1 (Experimental): liposomal doxorubicin: 40mg/m2 IV Day 1 every 28 days plus lenalidomide: 10 mg daily on Days 1-28 every 28 days
  Interventions: Drug: Lenalidomide; Drug: liposomal doxorubicin
- Phase I - Dose Level 2 (Experimental): liposomal doxorubicin: 40mg/m2 IV Day 1 every 28 days plus lenalidomide: 15 mg daily on Days 1-28 every 28 days
  Interventions: Drug: Lenalidomide; Drug: liposomal doxorubicin
- Phase 2 (Experimental): liposomal doxorubicin: 40mg/m2 IV Day 1 every 28 days plus lenalidomide: maximum tolerated dose from Phase I portion of the study (10mg) daily on Days 1-28 every 28 days
  Interventions: Drug: Lenalidomide; Drug: liposomal doxorubicin

INTERVENTIONS:
Drug: Lenalidomide — administered by mouth at the assigned dose daily for each 28 day cycle
  Other Names: Revlimid
Drug: liposomal doxorubicin — administered at a fixed dose of 40 mg/m^2 intravenously (IV) on day 1 of each 28 day cycle
  Other Names: Caelyx®

SUMMARY:
RATIONALE: Lenalidomide may stop the growth of cancer by blocking blood flow to the tumor. Drugs used in chemotherapy, such as doxorubicin hydrochloride liposome, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving lenalidomide together with doxorubicin hydrochloride liposome may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of lenalidomide when given together with doxorubicin hydrochloride liposome in treating patients with recurrent ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Phase I - Primary

* To determine the maximum tolerated dose of lenalidomide when combined with fixed dose pegylated liposomal doxorubicin hydrochloride in women with recurrent ovarian epithelial, fallopian tube, or primary peritoneal cancer.

Phase II - Define the best overall response induced by lenalidomide in recurrent ovarian cancer patients

Secondary

* To obtain preliminary information on toxicity, response, and time to progression (duration of response) of these patients.
* Progression free survival

Phase I OUTLINE: This is a dose-escalation study of lenalidomide. Patients receive oral lenalidomide once daily on days 1-28 and pegylated liposomal doxorubicin hydrochloride intravenously (IV) on day 1. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Phase II OUTLINE: The phase II component will include patients with measurable disease per Response Evaluation Criteria In Solid Tumors (RECIST) criteria treated at lenalidomide 10 mg days 1-28 days of a 28 day cycle (Maximum Tolerated Dose from phase I) with liposomal doxorubicin 40 mg/m^2 to determine efficacy and safety of the combination therapy. (Effective with April 2010 revision)

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer which has recurred or is resistant to prior treatment with at least one platinum based regimen and meeting at least one of the following criteria:

  * Platinum refractory - progression during the first six cycles of first line therapy with a platinum based regimen
  * Platinum resistant - progression within 6 months of completing first line platinum based chemotherapy
  * Platinum sensitive - progression more than 6 months of completing first line platinum based chemotherapy
  * Disease that has progressed while receiving or recurred within 6 months of completing platinum based second-line therapy Patients who have failed a second line therapy more than 6 months after completing treatment or have had more than 2 prior chemotherapy regimens will not be eligible for this study.
* Measurable disease per Response Evaluation Criteria In Solid Tumors (RECIST) criteria defined as one or more lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as > or = 20 mm with conventional techniques (CT, PET/CT, MRI, X-ray) or as > or = 10 mm with spiral CT scan.

Patients entering the study during the dose escalation component who do not meet the measurable disease requirement may enter with elevated CA 125 levels only if previously normal or stable CA 125 levels are documented after the completion of the prior chemotherapy regimen.

* Age > or = 18 years at the time of signing of consent form
* Gynecologic Oncology Group (GOG) performance status of < or = 2
* Laboratory test results within these ranges within 14 days prior to study registration:

  * Absolute neutrophil count > or = 1.5 x 10^9/L
  * Platelet count > or = 100 x 10^9/L
  * Serum creatinine < or = 1.5 mg/dL
  * Total bilirubin < 1.2 mg/dL
  * AST (SGOT) and ALT (SGPT) < or = 2 x upper limit of institutional normal (ULN) or < or = 5 x ULN if hepatic metastases are present.
* The left ventricular ejection fraction must be at or above the lower institutional limits of normal (as assessed by MUGA scan or echocardiogram) obtained within 28 days prior to registration.
* Peripheral neuropathy ≤ grade 2 (CTCAE v 3.0).
* Patients who are taking a stable or decreasing dose of concomitant systemic steroids during the study must agree to also take low dose aspirin and/or other platelet-active, anti-thrombotic medication (medication[s] used will be decided by the Investigator) while receiving study drug and for 30 days after study drug is discontinued.
* All previous cancer therapy, including chemotherapy, hormonal therapy and surgery, must have been discontinued at least 28 days prior to treatment in this study. Use of thalidomide, or structurally related compounds, radiation, or biologic response modifiers must be discontinued at least 2 weeks prior to treatment in this study.
* Progression free of prior malignancies for > or = 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin)
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

  * A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

Exclusion criteria:

* Histologic diagnosis of borderline or low malignant potential epithelial carcinoma.
* Any serious medical condition, laboratory abnormality, or psychiatric illness that, in the opinion of the investigator, would prevent the patient from signing the consent form.
* Prior history of myocardial infarction, congestive heart failure, or arrhythmia requiring medication. History of uncontrolled hypertension. History of systolic or diastolic dysfunction. EKG evidence of ventricular hypertrophy, conduction abnormality, or serious arrhythmia.
* History of deep vein thromboembolism (DVT) within the previous 6 months, history of thrombocytopenia or bleeding disorders.
* Pregnant or breast feeding females. Lenalidomide is pregnancy category X.
* Any condition, including the presence of laboratory abnormalities, which places the patient at unacceptable risk if she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 28 days of study registration.
* Known hypersensitivity reaction > grade 2 to thalidomide or structurally related compounds
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
* Any prior use of lenalidomide or liposomal doxorubicin
* Concurrent use of other anti-cancer agents or treatments
* Known positive for HIV or infectious hepatitis, type A, B or C
* Uncontrolled hyper- or hypo- calcemia, glycosemia or thyroidism

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Levi S. Downs, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Medical Center - Fairview, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Fifteen subjects were enrolled in this combined phase l/ll study - 11 subjects in phase l and 4 in phase ll. Six of the subjects enrolled in phase 1 were treated at the maximum tolerated dose (MTD) and their data was included in the phase 2 analysis as allowed by the protocol.
Groups:
- Phase 1 - Dose Level 2: liposomal doxorubicin: 40mg/m2 IV Day 1 every 28 days plus lenalidomide: 15 mg daily on Days 1-28 every 28 days
- Phase 2 - Dose Level 1: liposomal doxorubicin: 40mg/m2 IV Day 1 every 28 days plus lenalidomide: maximum tolerated dose from Phase I portion of the study (10mg) daily on Days 1-28 every 28 days
Period: Phase l
Arm/Group | Phase 1 - Dose Level 1 | Phase 1 - Dose Level 2 | Phase 2 - Dose Level 1
Started | 6 | 5 | 0
Completed | 6 | 5 | 0
Not Completed | 0 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1 - Dose Level 1 | Phase 1 - Dose Level 2 | Phase 2 - Dose Level 1
Started | 6 | 0 | 4
Completed | 6 | 0 | 3 (One participant was removed from the study after 2 weeks of treatment due to skin toxicity.)
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: One of the 4 subjects enrolled in the Phase 2 portion of the study was removed from the study 2 weeks after the start of treatment due to a skin rash leaving 9 evaluable subjects for the Phase 2 analysis. All 15 subjects from both the Phase 1 and Phase 2 portions of the trial were included in the Serious and Non-Serious Adverse Events analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 - Dose Level 1 | Phase 1 - Dose Level 2 | Phase 2 | Total
Number analyzed (Participants) | 6 | 5 | 4 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 9
  >=65 years | 3 | 2 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 4 | 15
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 4 | 15

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 - Maximum Tolerated Dose (MTD) of Lenalidomide When Combined With Fixed Dose Liposomal Doxorubicin in Women With Recurrent Epithelial Ovarian, Fallopian Tube, and Primary Peritoneal Cancer
Description: The maximum tolerated dose (MTD) reflects the highest dose of Lenalidomide when combined with fixed dose Liposomal Doxorubicin at which no more than one out of 6 participants experiences a dose limiting toxicity (DLT).
Time Frame: 1 cycle (28 days)
Measure: Number; unit: milligrams (mg)
Groups:
- Lenalidomide With Liposomal Doxorubicin: Patients treated with a combination of lenalidomide and liposomal doxorubicin for recurrent epithelia ovarian, fallopian tube or primary peritoneal cancer.
  Lenalidomide: Administered by mouth at the assigned dose; beginning at 10 mg and schedule of each 28 day cycle
  pegylated liposomal doxorubicin hydrochloride: Liposomal doxorubicin at a fixed dose of 40 mg/m^2 intravenously (IV) on day 1 of each 28 day cycle
Arm/Group | Lenalidomide With Liposomal Doxorubicin
Number analyzed (Participants) | 11
milligrams (mg) | 10

2. Primary Outcome: Phase 1 - Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: DLT is defined as the inability to complete cycle 1 and/or begin cycle 2 within 7 days of the planned start due to a grade 4 or greater hemtologic toxicity or a grade 3 or greater non-hematologic toxicity. Grading was based on Common Toxicity Criteria (CTC) Version 4.
Time Frame: within 5 weeks of starting treatment
Measure: Number; unit: participants
Arm/Group | Phase 1 - Dose Level 1 | Phase I - Dose Level 2 | Phase 2
Number analyzed (Participants) | 6 | 5 | 0
participants | 0 | 2 |

3. Primary Outcome: Phase 2 - Number of Subjects Achieving a Partial or Complete Response
Description: Partial response is defined as:
  At least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum longest diameter. To be assigned a status of partial response, changes in tumor measurements must be confirmed by repeat assessments performed no less than four weeks after the criteria for response are first met.
  Complete response is defined as:
  The disappearance of all target lesions. To be assigned a status of complete response, changes in tumor measurements must be confirmed by repeat assessments performed no less than four weeks after the criteria for response are first met.
Time Frame: 3 months after starting treatment
Measure: Number; unit: participants
Arm/Group | Phase 1 - Dose Level 1 | Phase I - Dose Level 2 | Phase 2
Number analyzed (Participants) | 0 | 0 | 9
participants |  |  | 1

4. Secondary Outcome: Phase 2 - Number of Subjects Who Are Progression-Free and Alive
Description: Progression is defined as:
  At least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of one or more new lesion(s).
Time Frame: 3 months after starting treatment
Measure: Number; unit: participants
Arm/Group | Lenalidomide With Liposomal Doxorubicin
Number analyzed (Participants) | 9
participants | 8

5. Secondary Outcome: Phase 2 - Number of Subjects Who Are Progression-Free and Alive
Description: Progression is defined as:
  At least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurement, or the appearance of one or more new lesion(s).
Time Frame: 6 months after starting treatment
Measure: Number; unit: participants
Groups:
- Lenalidomide With Liposomal Doxorubicin: Patients treated with a combination of lenalidomide and liposomal doxorubicin fpr recurrent epithelia ovarian, fallopian tube or primary peritoneal cancer.
  Lenalidomide: Administered by mouth at the assigned dose; beginning at 10 mg and schedule of each 28 day cycle
  pegylated liposomal doxorubicin hydrochloride: Liposomal doxorubicin at a fixed dose of 40 mg/m^2 intravenously (IV) on day 1 of each 28 day cycle
Arm/Group | Lenalidomide With Liposomal Doxorubicin
Number analyzed (Participants) | 9
participants | 5

ADVERSE EVENTS:
Groups:
- Phase 1 - Dose Level 1; Phase 2: Patients treated with a combination of lenalidomide and liposomal doxorubicin for recurrent epithelia ovarian, fallopian tube or primary peritoneal cancer.
  Lenalidomide: Administered by mouth at the assigned dose of 10 mg daily of each 28 day cycle
  pegylated liposomal doxorubicin hydrochloride: Liposomal doxorubicin at a fixed dose of 40 mg/m^2 intravenously (IV) on day 1 of each 28 day cycle
- Phase 1 - Dose Level 2: Patients treated with a combination of lenalidomide and liposomal doxorubicin for recurrent epithelia ovarian, fallopian tube or primary peritoneal cancer.
  Lenalidomide: Administered by mouth at the assigned dose of 15 mg daily of each 28 day cycle
  pegylated liposomal doxorubicin hydrochloride: Liposomal doxorubicin at a fixed dose of 40 mg/m^2 intravenously (IV) on day 1 of each 28 day cycle
Arm/Group | Phase 1 - Dose Level 1 | Phase 1 - Dose Level 2 | Phase 2
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/5 | 1/4
Other Adverse Events (participants affected / at risk) | 6/6 | 4/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 - Dose Level 1 (N=6) | Phase 1 - Dose Level 2 (N=5) | Phase 2 (N=4)
fever (General disorders) | 0 | 0 | 1 (1)
febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 (1) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 - Dose Level 1 (N=6) | Phase 1 - Dose Level 2 (N=5) | Phase 2 (N=4)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Blurred vision (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 2
Constipation (Gastrointestinal disorders) | 2 | 2 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1
Mucositis, oral (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 3
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Anal pain (Gastrointestinal disorders) | 0 | 1 | 0
Edema, limbs (General disorders) | 1 | 0 | 1
Fatigue (General disorders) | 2 | 3 | 2
Pain NOS (General disorders) | 0 | 0 | 2
Chills (General disorders) | 0 | 1 | 0
Bronchial infection (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 1 | 2
Platelet count decreased (Investigations) | 0 | 1 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle cramps, foot (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 2
Burning with urination, intermittent (Renal and urinary disorders) | 0 | 0 | 1
Bladder discomfort NOS (Renal and urinary disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Shortness of breath with intermittent wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Plantar palmar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculopapular (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Red spots, hands (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Infection, toe (Infections and infestations) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash, lower extremeities (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0
Phlebitis, arm (Vascular disorders) | 0 | 0 | 1
Hip pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No